CLINICAL TRIAL: NCT02338440
Title: Pharmacokinetic Study of Lipo-PGE1 for Prevention of VOD After HSCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUCH-HSCT-lipoPGE1
Record Dates: First submitted 2014-12-30; First posted 2015-01-14 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Veno-occlusive Disease; Child

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lipoprostaglandin E1 treatment arm (Experimental): * lipoprostaglandin E1 1mcg/kg/day, continuous infusion
  * lipoprostaglandin E1 1.5mcg/kg/day, continuous infusion (for patients with elevating total bilirubin, hepatomegaly, right upper quadrant abdominal pain, unexplained weight gain)
  Interventions: Drug: lipoprostaglandin E1

INTERVENTIONS:
Drug: lipoprostaglandin E1 — Blood sampling before administration (baseline), between 1 hour to 72 hours from administration (plateau 1), 72 hours after engraftment (plateau 2), when the clinician determine to do blood sampling because of change of kidney/liver function change (optional 1), 72 hours from the change of lipoprostaglandin E1 concentration change (optional 2)
  Other Names: Alostin

SUMMARY:
Veno-occlusive disease (VOD) after hematopoietic stem cell transplantation (HSCT) remains the major complication. VOD occurs in 11-31% of pediatric HSCT and the mortality reaches up to 50%.

Prostaglandin E1 (PGE1) have been reported to prevent and relieve the severity of VOD by Gluckman et al.. Lipo-PGE1 is a transporter of PGE1, which is superior in concentrating PGE1 and acts for prolonged time. Because of the prolonged effective time, lipo-PGE1 acts comparable effects by 1/4~1/8 of PGE1 dose. Empirically, pediatric HSCT centers adopt lipo-PGE1 in dose of 1 mcg/kg/day (0.042 mcg/kg/hr), which is 1/7 of the dose recommended by Gluckman, et al. This prospective study will investigate the concentration of lipo-PGE1 with preventive lipo-PGE1 with empirical dose (1 mcg/kg/day).

DETAILED DESCRIPTION:
Primary Objective: To evaluate the pharmacokinetics of lipo-PGE1. Secondary objective: To evaluate the relation between lipo-PGE1 concentration and VOD occurrence, severity.

Inclusion criteria

1. Patients undergoing HSCT with high risk of VOD who cannot use low dose heparin.

   * high risk of VOD : previous radiotherapy, liver function abnormality, children, conditioning regimen including busulfan or total body irradiation
   * contraindication of heparin : low platelet count, bleeding tendency, allergy
2. Patients (or one of parents if patients age < 19) should sign informed consent.

Exclusion criteria

1. Patient with heart failure.
2. Patient with bleeding (intracranial hemorrhage, gastrointestinal tract bleeding, hemoptysis).
3. History of hypersensitivity reaction as shock to lipo-PGE1.
4. Psychiatric disorder that would preclude compliance.
5. If the clinician decides that there is a condition improper for the clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing HSCT with high risk of VOD who cannot use low dose heparin.

   * high risk of VOD : previous radiotherapy, liver function abnormality, children, conditioning regimen including busulfan or total body irradiation
   * contraindication of heparin : low platelet count, bleeding tendency, allergy
2. Patients (or one of parents if patients age < 19) should sign informed consent.

Exclusion Criteria:

1. Patient with heart failure.
2. Patient with bleeding (intracranial hemorrhage, gastrointestinal tract bleeding, hemoptysis).
3. History of hypersensitivity reaction as shock to lipo-PGE1.
4. Psychiatric disorder that would preclude compliance.
5. If the clinician decides that there is a condition improper for the clinical study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
pharmacokinetics of lipo-PGE1 (Lipo-PGE1 level (B, P1, P2, O1, O2)) | baseline (pre-dose), 1 to 72 hours from starting continuous infusion of lipo-PGE1
  Lipo-PGE1 drug level of time points (B, P1, P2, O1, O2)

SECONDARY OUTCOMES:
Incidence of VOD after transplantation | until 3 months after transplantation
  cumulative incidence of VOD until 3 months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, MD, PhD, Principal Investigator — Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, Chongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided